CLINICAL TRIAL: NCT02293044
Title: A Pilot Clinical Study to Evaluate the Safety and Efficacy of a Self-Applied Oxalate Strip on Adjacent Teeth With Dentinal Hypersensitivity
Brief Title: A Study to Evaluate the Safety and Efficacy of an Oxalate Strip on Adjacent Teeth With Dentinal Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014115
Record Dates: First submitted 2014-11-07; First posted 2014-11-18 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Dentin Sensitivity
Keywords: Sensitivity
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity

ARMS (1):
- Crest® Sensi-Stop™ Strips (Experimental): Self Applied
  Interventions: Device: Crest® Sensi-Stop™ Strips

INTERVENTIONS:
Device: Crest® Sensi-Stop™ Strips

SUMMARY:
This study will compare the safety and effectiveness of a potassium oxalate desensitizer on adjacent teeth with dentinal hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* sign an informed consent form and be given a copy
* be in good general health as determined by the Investigator/designee
* have at least one pair of adjacent teeth, each of which has a screening score of - -greater than or equal to 1 on the Schiff Sensitivity Scale in response to the cold water challenge.

Exclusion Criteria:

* severe periodontal disease, as characterized by purulent exudate, generalized mobility, and/or severe recession
* active treatment for periodontitis
* any diseases or conditions that might interfere with the subject safely completing the study
* inability to undergo study procedures
* fixed facial orthodontic appliances
* self-reported pregnancy or nursing
* a history of kidney stones
* known allergies to the following ingredients; aqua, glycerin, cellulose gum, dipotassium oxalate, carbomer, sodium hydroxide, sodium benzoate, and potassium sorbate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Gerlach, DDS, MPH, Principal Investigator — Procter and Gamble
Locations (1):
- Oral Health Science Center, Mason, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Crest® Sensi-Stop™ Strips: Self Applied
  Crest® Sensi-Stop™ Strips
Period: Overall Study
Arm/Group | Crest® Sensi-Stop™ Strips
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Fifteen (15) subjects received study products. Fifteen (15) subjects completed the study.
Arm/Group | Crest® Sensi-Stop™ Strips
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 2
  Ethnicity: Black | 1
  Ethnicity: Caucasian | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Cold Water Challenge
Description: The Schiff Sensitivity Scale was assessed for each test tooth via a cold water challenge. The examiner recorded the Schiff Index score corresponding to the response to the cold water challenge. The Schiff Index Sensitivity scale is scored as follows- 0: tooth/subject did not respond to stimulus, 1: tooth/subject responds to stimulus, but does not request discontinuation of stimulus, 2: tooth/subject responds to stimulus and requests discontinuation or moves form stimulus, 3: tooth/subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A negative change from Baseline score represents a decrease in sensitivity from baseline. The mean change from Baseline was calculated for this measure.
Time Frame: 1 Day
Population: Fifteen (15) subjects received study products. Fifteen (15) subjects completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crest® Sensi-Stop™ Strips
Number analyzed (Participants) | 15
Units on a scale | -1.00 (0.76)

2. Secondary Outcome: Change From Baseline Visual Analog Scale
Description: Visual Analog Scale (VAS) - subjects are asked to look at a VAS and designate the level of hypersensitivity they experienced as a result of the thermal and water challenges using a continuum scale of 0 = No tooth pain up to 100 = Worst tooth pain ever experienced. A negative change from Baseline score represents a decrease in sensitivity from baseline. The mean change from Baseline was calculated for this measure.
Time Frame: 1 Day
Population: Fifteen (15) subjects received study products. Fifteen (15) subjects completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crest® Sensi-Stop™ Strips
Number analyzed (Participants) | 15
Units on a scale | -18.00 (13.61)

ADVERSE EVENTS:
Arm/Group | Crest® Sensi-Stop™ Strips
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes